CLINICAL TRIAL: NCT02429375
Title: Phase IB/II Study of Mocetinostat (MGCD0103) Plus Brentuximab Vedotin (SGN-35) in Patients With Relapsed or Refractory Hodgkin Lymphoma
Brief Title: Mocetinostat (MGCD0103) Plus Brentuximab Vedotin (SGN-35) in Patients With Relapsed or Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: MethylGene Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-232
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Results first posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-03

CONDITIONS: Hodgkin Lymphoma
Keywords: Mocetinostat (MGCD0103); Brentuximab Vedotin (SGN-35); Relapsed; Refractory
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — mocetinostat; Brentuximab Vedotin

ARMS (1):
- Mocetinostat (MGCD0103) Plus Brentuximab Vedotin (SGN-35) (Experimental): Patients with relapsed or refractory Hodgkin lymphoma will receive brentuximab vedotin combined with mocetinostat. For the phase I portion of the study, patients will be enrolled in a traditional 3 + 3 phase 1 design on sequential dosing cohorts in order to determine the maximum tolerated dose (MTD) of mocetinostat when given with brentuximab vedotin. Once the MTD is determined, (up to) an additional 26 patients will be enrolled on to the phase II portion of the study at the MTD to determine the response rate and toxicity associated with treatment. The phase Ib and II study will include a lead-in with mocetinostat alone for 1 week followed by the combined treatment beginning day 15 following initiation of mocetinostat.
  Interventions: Drug: Mocetinostat Plus Brentuximab Vedotin

INTERVENTIONS:
Drug: Mocetinostat Plus Brentuximab Vedotin — All patients will receive a 1-week lead-in with mocetinostat alone (administered days 1, 3, and 5). Patients with palpable peripheral lymph nodes will undergo FNA before and after this 1 week treatment. Cycle 1 will then begin 15 days (+/-3 days) following initiation of the lead-in.
  Other Names: MGCD0103; SGN-35

SUMMARY:
The purpose of this study is to find out how safe and effective treatment with a new combination of drugs, mocetinostat and brentuximab vedotin, is in treating cancer. There will be 2 parts to this trial: a phase I part and a phase II part.

Brentuximab vedotin is approved by the U.S. Food and Drug Administration (FDA) to be given to patients with Hodgkin Lymphoma. Mocetinostat is an experimental drug that has been given to patients with Hodgkin lymphoma in another clinical trial. When given alone, mocetinostat caused lymphoma to shrink in about 1 out of 4 patients with Hodgkin lymphoma. This is the first study that will give mocetinostat and brentuximab vedotin together.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed CD30 positive relapsed or refractory Hodgkin lymphoma
* Measurable disease, as defined by the International Harmonization Project.14
* Patients must have failed autologous stem cell transplant or at least 2 prior cytotoxic regimens for Hodgkin lymphoma. Patients who have failed only 1 prior cytotoxic regimen for Hodgkin lymphoma are permitted to enroll as long as they are not eligible for autologous stem cell transplant.
* Age ≥18
* ECOG performance status ≤2 (Karnofsky ≥60%)
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,000/mcL
  * platelets ≥75,000/mcL
  * total bilirubin within normal institutional limits or < 3x the upper limit of normal in patients with Gilbert's disease
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * Creatinine ≤1.5 x institutional upper limit of normal OR creatinine clearance ≥40 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* QTc ≤ 500 ms
* The effects of mocetinostat and brentuximab vedotin on the developing human fetus are potentially harmful. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of mocetinostat and brentuximab vedotin administration.
* Patients with known HIV infection must have CD4 count greater than 200.

Exclusion Criteria:

* Presence of a small (or greater size) pericardial effusion; definitions of pericardial effusions by echocardiographic assessment.
* Patients who have had chemotherapy or radiotherapy within 3 weeks prior to entering the study
* Patients who have not recovered from adverse events due to agents administered more than 3 weeks earlier.
* Patients who are receiving any other investigational agents.
* Patients with known cerebral or meningeal involvement by lymphoma are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to mocetinostat or brentuximab vedotin.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled diabetes, clinically significant pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant or breastfeeding
* Previous primary progression or grade 3 toxicity on treatment with brentuximab vedotin
* Systemic steroids are allowed as long as they are tapered to the equivalent of 20mg prednisone daily or less by the start of cycle 2.
* Platelet or packed red blood cell transfusion within 14 days of pre-treatment evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-04-22 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 50mg Mocetinostat; Dose Level 2: 70mg Mocetinostat; Dose Level 3: 90mg Mocetinostat: Mocetinostat Plus Brentuximab Vedotin: All patients will receive a 1-week lead-in with mocetinostat alone (administered days 1, 3, and 5). Patients with palpable peripheral lymph nodes will undergo FNA before and after this 1 week treatment. Cycle 1 will then begin 15 days (+/-3 days) following initiation of the lead-in.
Period: Overall Study
Arm/Group | Dose Level 1: 50mg Mocetinostat | Dose Level 2: 70mg Mocetinostat | Dose Level 3: 90mg Mocetinostat
Started | 3 | 3 | 1
Completed | 3 | 3 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with relapsed or refractory Hodgkin lymphoma
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: 50mg Mocetinostat | Dose Level 2: 70mg Mocetinostat | Dose Level 3: 90mg Mocetinostat | Total
Number analyzed (Participants) | 3 | 3 | 1 | 7
Age, Continuous [Median (Full Range); unit: years] | 43 [24 to 62] | 30 [25 to 33] | 43 [43 to 43] | 33 [24 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 0 | 4
  Male | 2 | 0 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 2 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 1 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: For this objective the standard 3+3 dose-escalation scheme will be used. Patients will be accrued to the study in cohorts of 3 (starting with dose level 1). For any given dose an initial cohort of 3 patients will be treated at that dose. The dose level will be escalated if none of the 3 patients exhibits any DLT
Time Frame: 1 year
Population: Data were not collected
Groups:
- Mocetinostat (MGCD0103) Plus Brentuximab Vedotin (SGN-35): Patients with relapsed or refractory Hodgkin lymphoma will receive brentuximab vedotin combined with mocetinostat.
Arm/Group | Mocetinostat (MGCD0103) Plus Brentuximab Vedotin (SGN-35)
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 50mg Mocetinostat | Dose Level 2: 70mg Mocetinostat | Dose Level 3: 90mg Mocetinostat
Number analyzed (Participants) | 3 | 3 | 1
Participants
  Progression of Disease | 2 | 0 | 1
  Partial Response | 0 | 2 | 0
  Stable Disease | 0 | 1 | 0
  NA - Patient Withdrawal of Consent | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dose Level 1: 50mg Mocetinostat | Dose Level 2: 70mg Mocetinostat | Dose Level 3: 90mg Mocetinostat
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: 50mg Mocetinostat (N=3) | Dose Level 2: 70mg Mocetinostat (N=3) | Dose Level 3: 90mg Mocetinostat (N=1)
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: 50mg Mocetinostat (N=3) | Dose Level 2: 70mg Mocetinostat (N=3) | Dose Level 3: 90mg Mocetinostat (N=1)
White blood cell decreased (Investigations) | 0 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Cholesterol high (Investigations) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
INR increased (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT02429375/Prot_SAP_000.pdf